CLINICAL TRIAL: NCT00281567
Title: A Randomised, Double-blind, Double-dummy, Placebo-controlled, Crossover Efficacy and Safety Comparison of 4-week Treatment Periods of Two Doses [5 μg (2 Actuations of 2.5 μg) and 10 μg (2 Actuations of 5 μg)] of Tiotropium Inhalation Solution Delivered by the Respimat Inhaler, Tiotropium Inhalation Powder Capsule (18μg) Delivered by the HandiHaler in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety Comparison of Tiotropium Inhalation Solution (Respimat Inhaler) and Spiriva HandiHaler in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205.250
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: Tiotropium
Device: Respimat SMI
Device: HandiHaler

SUMMARY:
Comparison of lung function response between tiotropium inhalation solution and Spiriva HandiHaler.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* FEV1 < 60% predicted
* FEV1 < 70% of FVC
* Smoking history of 10 pack-years

Exclusion Criteria:

* Significant other disease than COPD
* Recent history of MI (1 year or less)
* Cardiac arrhythmia requiring drug therapy
* History of asthma, allergic rhinitis or eosinophil count > 600 mm3
* Symptomatic prostatic hypertrophy or bladder neck obstruction
* Known narrow-angle glaucoma
* Abnormal baseline hematology, blood chemistry or urinalysis
* History of cancer within last 5 years
* Life-threatening pulmonary obstruction
* Cystic fibrosis or bronchiectasis
* Tuberculosis
* Pulmonary resection

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2002-08; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Comparison of trough FEV1 values at the end of 4-week treatment with tiotropium inhalation solution (5 mcg, 10 mcg) to that achieved with tiotropium inhalation powder (Spiriva 18 mcg).

SECONDARY OUTCOMES:
Trough forced vital capacity (FVC) response after 4 weeks (change from baseline) | baseline until week 28
Peak response (FEV1 and FVC) to first dose | within 3 hours to first dose
Peak response (FEV1 and FVC) after 4 weeks | within 3 hours after 4 weeks
FEV1 AUC0-12h and FVC AUC0-12h response after 4 weeks | after 4 weeks
FEV1 AUC0-3h and FVC AUC0-3h response after the first dose and after 4 weeks | after first dose and after 4 weeks
Individual FEV1and FVC measurements at each time point | up to 28 weeks
Pre-dose morning and evening peak expiratory flow rate (PEFR) measured by patients | up to 28 weeks
Number of occasions of rescue therapy used as required (p.r.n. salbutamol) | up to 28 weeks
Median time to onset of therapeutic response after first dose | after 4 weeks
Number of patients with 15% response above baseline for each treatment at each timepoint after first dose | at week 4, 12, 20
Number of patients with 15% response above baseline for each treatment at each timepoint after 4 weeks | at week 8, 16, 24

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim KG
Locations (2):
- Boehringer Ingelheim Investigational Site, Study Chairs Or Principal Investigators, Belgium
- Boehringer Ingelheim Investigational Site, Study Chairs Or Principal Investigators, Netherlands